CLINICAL TRIAL: NCT07337395
Title: Identification of Proteomic Changes in Patients With Generalized Myasthenia Gravis Treated With Ravulizumab: Insights Into Neuromuscular Junction Regeneration
Brief Title: Proteomic Changes in Patients With Myasthenia Gravis and Ravulizumab
Acronym: PROMPT
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 8167
Record Dates: First submitted 2025-12-19; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Myasthenia Gravis Generalised
Keywords: Myasthenia Gravis; Ravulizumab; Proteomic changes
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

SUMMARY:
Myasthenia gravis (MG) is an autoimmune neuromuscular disorder primarily caused by antibodies targeting postsynaptic components of the neuromuscular junction, most commonly the acetylcholine receptor (AChR). In AChR-positive generalized MG, IgG1 and IgG3 antibodies activate the classical complement pathway, leading to membrane attack complex-mediated damage of the postsynaptic membrane and impaired neuromuscular transmission. Complement inhibition has therefore emerged as an effective therapeutic strategy.

Ravulizumab, a long-acting monoclonal antibody targeting complement component C5, has demonstrated clinical efficacy in reducing disease severity in patients with AChR-positive generalized MG. However, clinical responses to complement inhibition remain heterogeneous, and reliable biomarkers to monitor treatment response and neuromuscular junction recovery are currently lacking.

Blood-based proteomics represents a powerful approach for identifying molecular changes associated with disease activity and treatment response. In particular, aptamer-based proteomic platforms such as the SomaScan® assay allow high-throughput, highly sensitive quantification of thousands of circulating proteins from small volumes of plasma or serum.

The primary aim of this study is to identify proteomic changes in patients with generalized MG treated with Ravulizumab, with a specific focus on proteins involved in neuromuscular junction regeneration and repair. By leveraging advanced proteomic technologies in a real-world clinical setting, this study seeks to identify biomarkers that may help monitor treatment response, guide optimization of concomitant immunosuppressive therapies, and improve patient stratification. Ultimately, the identification of molecular pathways associated with neuromuscular junction regeneration may open new therapeutic perspectives for autoimmune neuromuscular disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Diagnosis of generalized anti-AChR positive Myasthenia Gravis;
* Need for therapy with Ravulizumab drugs according to the therapeutic indications approved by AIFA;
* Signed informed consent to the study.

Exclusion Criteria:

* Age <18 years;
* Concomitant autoimmune diseases;
* Insufficient availability of clinical information;
* Ongoing neoplasia or infection at the time of biological sample collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with generalized Myasthenia Gravis positive for anti-AChR antibodies undergoing therapy with Ravulizumab
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
To identify significant changes in plasma protein profiles in patients with generalized myasthenia gravis (gMG) treated with Ravulizumab. | 26 weeks
  To identify changes in plasma proteins after 10 and 26 weeks of treatment with Ravulizumab compared with baseline, using proteomic technology.

SECONDARY OUTCOMES:
To identify plasma proteins associated with a clinically meaningful improvement in patients with gMG. | 26 weeks
  To analyze correlations between plasma protein profiles and clinical outcome measures in patients with gMG after 10 and 26 weeks of treatment with Ravulizumab.
To identify potential biomarkers of neuromuscular junction regeneration in patients with gMG. | 24 months
  To create a dedicated database and perform a literature review to determine whether any of these proteins may represent potential biomarkers of neuromuscular junction regeneration in patients with gMG.

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Iorio, Prof, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy